CLINICAL TRIAL: NCT00580697
Title: Prevalence of Lower Urinary Tract Symptoms in Women With Gynecologic Malignancy Planning to Undergo Surgical Management
Status: Withdrawn | Type: Observational
Why Stopped: Nonapplicable clinical trial
Sponsor: University of California, Irvine (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-4825
Record Dates: First submitted 2007-12-19; First posted 2007-12-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Lower Urinary Tract Symptoms; Gynecologic Malignancy
Keywords: Lower urinary tract symptoms; Gynecologic malignancy; Urinary incontinence; Fecal incontinence; Frequency; Voiding dysfunction; Sexual dysfunction
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence; Fecal Incontinence; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is to determine the prevalence of lower urinary tract symptoms in women undergoing surgery for gynecologic malignancy.

DETAILED DESCRIPTION:
Lower urinary tract symptoms, including urinary incontinence, voiding dysfunction, urgency, frequency, fecal incontinence, as well as sexual dysfunction, is directly affected by gynecologic malignancies and the surgical and medical management of those malignancies. Increased risk of injury to the urinary tract is a recognized complication of surgical and medical therapy of gynecologic malignancies. To date, only a few studies have looked at the incidence of lower urinary tract symptoms at the time of diagnosis of gynecologic malignancy and prior to treatment, and there have been no published studies describing the incidence of sexual dysfunction at the time of diagnosis and prior to therapy of gynecologic malignancies. However, sexual dysfunction has been described in patients with urinary incontinence and pelvic organ prolapse and following surgery for incontinence and pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a new diagnosis of gynecologic malignancy who plan to undergo surgical management, including cervical, endometrial, and ovarian cancer.

Exclusion Criteria:

* Subjects less than 18 years of age
* Subjects unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Have a diagnosis of a gynecologic malignancy: cervical, endometrial, or ovarian cancer, and plan to have surgry for the cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The outcome will be measured using validated general and condition-specific questionnaires. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Noblett, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States